CLINICAL TRIAL: NCT04924452
Title: Efficiency of Er:YAG Laser Therapy in Combination With Behaviour Management Technique in Reducing Anxiety Among Paediatric Dental Patients
Brief Title: Er:YAG Laser Therapy in Combination With Behaviour Management Technique in Reducing Anxiety Among Paediatric Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Plovdiv Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MedicalUniversity_BMT
Record Dates: First submitted 2021-06-03; First posted 2021-06-14 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Dental Caries; Dental Anxiety; Behavior
Keywords: Er:YAG laser; anxiety; management technique; paediatric dentistry
MeSH Terms: conditions — Dental Caries; Behavior; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: randomized parallel-group controlled clinical study
Who Masked: Participant
Masking Description: The randomisation will be independent and the patients and parents/guardians will remain blinded to group status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Er:YAG laser therapy (Experimental): Er:YAG laser will be used for enamel conditioning of the occlusal surfaces of the permanent molars before sealant application as well as the standardized caries treatment.
  Interventions: Procedure: Laser conditioning and Sealant application; Device: Er:YAG laser therapy
- Conventional therapy (Active Comparator): Conventional rotary instruments will be used for caries treatment.
  Interventions: Procedure: Sealant application; Procedure: Conventional therapy

INTERVENTIONS:
Procedure: Laser conditioning and Sealant application — Sealant application protocol includes: a low-speed rubber cup and pumice paste (CleanPolish, Kerr) will be used for 30 seconds for cleaning and polishing of the occlusal surface of the chosen permanent molar; tooth surface will be washed for debris and organic residue removal and dried with air spray; isolation; laser conditioning of the occlusal enamel surface. The parameter settings used will be: tip-to-tissue distance 1.5mm from the tooth surface; tip diameter 600 µm; laser energy 70 mJ; pulse frequency 10 Hz; water spray level 8; average power 0.7 W; energy density 67 J/cm2; tooth surface will be etched with 35% phosphoric acid gel (Etching gel, DMP Ltd) for 30 seconds and rinsed for the same time; reisolation; tooth surface will be dried with air spray for 15s; fissure sealant application (Pit&Fissure Sealant, DMP Ltd); light cured for 20 seconds.
  Arms: Er:YAG laser therapy
Procedure: Sealant application — Sealant application protocol includes: a low-speed rubber cup and pumice paste (CleanPolish, Kerr) will be used for 30 seconds for cleaning and polishing of the occlusal surface of the chosen permanent molar; tooth surface will be washed for debris and organic residue removal and dried with air spray; isolation; tooth surface will be etched with 35% phosphoric acid gel (Etching gel, DMP Ltd) for 30 seconds and rinsed for the same time; reisolation; tooth surface will be dried with air spray for 15s; fissure sealant application (Pit&Fissure Sealant, DMP Ltd); light cured for 20 seconds.
  Arms: Conventional therapy
Device: Er:YAG laser therapy — Er:YAG laser (LiteTouch, Light Instruments LTD), emission wavelength 2940 nm will be used for caries removal - parameters: enamel removal - energy 100-200mJ; density 9.84-13.03 J/cm2, pulse frequency 20Hz; tip diameter 800 μm; water spray level 8; tip-to-tissue distance 0.5÷1 mm form the tooth surface; dentin removal - energy 100mJ; density 9.84 J/cm2, pulse frequency 20Hz; tip diameter 800 μm; water spray level 8; tip-to-tissue distance 0.5÷1 mm form the tooth surface. Restoration with compomer.
  Arms: Er:YAG laser therapy
Procedure: Conventional therapy — Conventional rotary instruments will be used for caries removal - high-speed and low-speed dental handpieces. Restoration with compomer.
  Arms: Conventional therapy

SUMMARY:
The aim of the study is to assess the efficacy of a modified version of the behaviour management technique Latent inhibition in combination with Er:YAG laser for achieving reduction of dental anxiety in paediatric dental patients. The main objectives are to compare dental anxiety felt during the laser and conventional dental treatment. The outcomes will be dental anxiety assessment by a self-reported anxiety during treatment in both group as well as measurement of heart rate dynamics during the procedures.

DETAILED DESCRIPTION:
When providing dental care to child patients with a high level of dental anxiety, the range of approaches are divided into two sections - use of behavior management techniques and application of alternative methods for caries removal. In attempt to reduce dental anxiety, they can be mixed and matched in accordance with the dentists' choice. Owing to the promoted advantages Er:YAG laser turns into an ideal alternative technique for hard dental tissue therapy in anxious pediatric patients.This is a protocol for a randomized controlled clinical trial. The participants will be children aged aged 6-12 years, requiring conservative treatment of occlusal carious lesions on a second primary molar. Patients will be randomly assigned to experimental or control group via computer-generated sequence. In both groups Latent inhibition will be used as an anxiety-management technique. In the experimental group caries treatment will be performed with Erbium:YAG laser, whereas in the control group with the conventional rotary instruments. Outcome measures will be dental anxiety felt before and after the treatment and the dynamics of heart rate, registered during the treatment session.

ELIGIBILITY:
Inclusion Criteria:

1. Participants in the study are children aged 6-12 years, compliant with the cognitive development of the child and the requirement for complete root development;
2. Children, requiring conservative treatment of occlusal carious lesions on a second primary molar, without spontaneous unprovoked pain, percussion or palpation pain or other symptoms, indicating pulp involvement or periodontal pathology. Lesions are classified as distinct cavity with visible dentin without prior restoration or sealants by the International Caries Detection and Assessment System (ICDAS) with code 05. Included are caries lesions only on vital teeth.
3. Children with one or more permanent molars giving indications for pit and fissure sealing;
4. Patients without previous experience with laser treatment of carious lesions;
5. Children who are not considered medically compromised or medically complex patients;
6. Verbal assent from the child willing to comply with all study procedures and protocol;
7. Obtained written informed consent by the patient's parent/guardian for participation in the study

Exclusion Criteria:

1. Patients who were undergoing therapy with neurological, sedative, analgesic, and/or anti-inflammatory drugs 7 days prior to treatment that might affect heart rate;
2. Children, who were first-time dental patients;
3. Children with systemic diseases or physiological development delays;
4. Children with mental or cognitive problems;
5. Present infectious diseases such as influenza, scarlet fever, etc.
6. Excluded are molars which are affected by disturbances in the development of dental structures (hypoplasia, hypomineralization, fluorosis)

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 82 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
self-report dental anxiety on a modified version of the self-report Faces Scale by LeBaron | Immediately after the dental treatment
  The scale comprises a row of five faces ranging from 'relaxed' to 'very worried' in combination with a visual analog scale of 0 - 10. Each child was asked to point to the face or choose the number which most closely depicted its state of anxiety.

SECONDARY OUTCOMES:
Heart rate | start: in the waiting room, at least 5 minutes before the dental treatment. End: at least 5 minutes after the dental treatment.
  Dynamics of heart rate, registered during the treatment session measured throughout the whole treatment session with a mobile pulse oximeter, placed on the index finger of the left hand

CONTACTS AND LOCATIONS:
Overall Officials: Maria Shindova, PhD, Principal Investigator — Medical University Plovdiv, Bulgaria
Locations (1):
- Department of Paediatric Dentistry, Faculty of Dental Medicine, Medical University - Plovdiv, Bulgaria, Plovdiv, Bulgaria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Belcheva A, Shindova M. Efficiency of ER:YAG laser therapy in combination with behaviour management technique in reducing anxiety among paediatric dental patients - a study protocol for a randomised clinical trial. BMJ Open. 2022 Sep 5;12(9):e054523. doi: 10.1136/bmjopen-2021-054523. PMID 36691137